CLINICAL TRIAL: NCT01912404
Title: A Placebo-Controlled, Multicenter, Double-Blind, Randomized Trial of IDN-6556 in Patients With Severe Alcoholic Hepatitis and Contraindications to Corticosteroid Therapy
Brief Title: Study of IDN-6556 in Patients With Severe Alcoholic Hepatitis and Contraindications to Steroid Therapy
Acronym: AH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to concern for high systemic drug levels that could exceed levels in toxicology studies.
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDN-6556-04; 5U01AA021788 (NIH)
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Alcoholic Hepatitis
Keywords: alcoholic hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IDN-6556 (Experimental): IDN-6556 capsules, 25 mg BID
  Interventions: Drug: IDN-6556
- Placebo (Placebo Comparator): Placebo capsules BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IDN-6556 — 25 mg BID for 28 days
  Other Names: emricasan; PF-03491390
  Arms: IDN-6556
Drug: Placebo — Placebo controlled
  Arms: Placebo

SUMMARY:
The main purpose of the study is to test if taking a study drug called emricasan (also known as IDN-6556 and PF-03491390) will affect overall patient survival after one month of treatment.

DETAILED DESCRIPTION:
The study will also see if overall patient survival is affected at 6 months, and if the study drug improves liver function.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent (either from patient or patient's legally acceptable representative), and understand and willing to comply with the requirements of the study
2. Male or female patients 21 years of age or older
3. Patients with alcoholic hepatitis defined as:

   1. History of heavy alcohol abuse use: >40 g/day in females and >60 g/day in males for most days in a minimum period of 6 months
   2. Consumed alcohol within 6 weeks of entry into the study
   3. Biochemical parameters of severe disease as evidenced by MELD score >20 but <35, or MELD score 35-40 if the SOFA score is <10
4. Willingness to utilize 2 reliable forms of contraception (for both males and females of childbearing potential) from screening to 1 month after the completion of study treatment
5. Patients with established contraindications to steroid use including but not limited to the following:

   1. GI bleed
   2. Active infection, including spontaneous bacterial peritonitis, based on positive blood culture, urine culture, or chest x-ray (if positive, must have been on antibiotics for at least 24 hours prior to study entry)
   3. Acute pancreatitis (increased lipase > 3x ULN or radiologic evidence)
   4. Positivity for hepatitis B (HBsAg+) or C virus (HCV+), and
   5. Renal failure

Exclusion Criteria:

1. Other or concomitant cause of liver disease as a result of:

   1. Autoimmune liver disease (positive anti-mitochondrial antibody and smooth muscle antibody, positive reading on anti-nuclear antibody titer >1:160)
   2. Metabolic liver disease (abnormal ceruloplasmin levels)
   3. Vascular liver disease
   4. Drug induced liver disease Note: Concurrent viral hepatitis is not excluded.
2. Co-infection with human immunodeficiency virus (HIV)
3. Sepsis as evidenced by positive blood or urine culture, or pneumonia as confirmed by x-ray
4. History of renal transplant and/or on dialysis at time of entry into study
5. Inflammatory bowel disease
6. Diagnosed or suspected systemic lupus erythematosus (SLE) and/or rheumatoid arthritis (RA)
7. Hepatocellular carcinoma (HCC) at entry into the study
8. Active non-liver malignancies other than curatively treated skin cancer (basal cell or squamous cell carcinomas)
9. Active tuberculosis on chest x-ray at study entry
10. History or presence of clinically concerning cardiac arrhythmias, or prolongation of screening (pre-treatment) QT or QTc interval of >480 milliseconds (msec)
11. Significant systemic or major illness other than liver disease, including coronary artery disease, cerebrovascular disease, pulmonary disease, renal failure, serious psychiatric disease, that, in the opinion of the Investigator would preclude the patient from participating in and completing the study
12. Patients requiring the use of vasopressors or inotropic support
13. Liver biopsy, if carried out, showing findings not compatible with alcoholic hepatitis
14. Any patient that has received any investigational drug or device within 30 days of dosing or who is scheduled to receive another investigational drug or device in the course of the study Note: Investigational drug includes any drug that is used off-label.
15. If female, known pregnancy, or has a positive urine or serum pregnancy test, or lactating/breastfeeding
16. If male, if partner is known to be pregnant at time of entry into study or becomes pregnant while patient is on study drug or up to 1 month after completion of study drug
17. Appropriate candidate for corticosteroid therapy
18. Treatment for alcohol hepatitis within 1 month of study entry with use of corticosteroids for >1 week or corticosteroid use at the time of entry into the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hagerty, MD, Study Director — Conatus Pharmaceuticals Inc.
Locations (3):
- United States (3):
  - Indiana University, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
Study was terminated early with insufficient subjects for meaningful analysis.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a placebo-controlled, double-blind, multicenter Phase 2 study in patients with alcoholic hepatitis who were contraindicated to receive corticosteroid therapy. The study consisted of a 7-day screening phase, a 28-day treatment phase, and a follow-up of 5 months. Total study duration for a patient was about 6 months.
Pre-assignment Details: Eligible patients were randomized in a 2:1 ratio to IDN-6556 25 mg or placebo administered twice daily for 28 days. During the treatment phase, the patients were assessed for safety and efficacy. Following the treatment phase, the patients were asked to return for follow-up visits at 1, 2, and 5 months after completion of study drug treatment.
Groups:
- IDN-6556: IDN-6556 capsules, 25 mg twice daily for 28 days
- Placebo: Matching Placebo capsules twice daily for 28 days
Period: Overall Study
Arm/Group | IDN-6556 | Placebo
Started | 3 | 2
Completed | 2 | 2
Not Completed | 1 | 0
Not completed — Due to personal reasons | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study in patients with alcoholic hepatitis who were contraindicated to receive corticosteroid therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDN-6556 | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (4.93) | 31 (1.41) | 41.6 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Survival
Time Frame: 28 days
Population: The study was prematurely stopped due to emerging data from another study showing ~10 to 12-fold higher exposures in patients with severe hepatic impairment compared to those with normal liver function. Since subjects with alcoholic hepatitis would likely have severe hepatic impairment, the study was stopped and survival data was not collected.
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | IDN-6556 | Placebo
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDN-6556 (N=3) | Placebo (N=2)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDN-6556 (N=3) | Placebo (N=2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (4)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Since the study was stopped early, no conclusions regarding efficacy can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less